CLINICAL TRIAL: NCT03055000
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study in Healthy Volunteers to Evaluate the Safety and Immunogenicity of AGS-v, a Universal Mosquito-Borne Disease Vaccine
Brief Title: Safety and Immunogenicity of a First-in-Human Mosquito Saliva Peptide Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 170059; 17-I-0059 (Other: NIAID)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2018-12

CONDITIONS: Mosquito-Borne Disease
Keywords: Mosquito-Borne Diseases; Universal Mosquito Vaccine; Mosquito Transmission; Vector Borne Viruses; Vaccine
MeSH Terms: conditions — Mosquito-Borne Diseases | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AGS-v (Experimental): AGS-v (unadjuvanted) as a suspension in WFI (0.5mL) on Day 0 and on Day 21
  Interventions: Biological: AGS-v
- AGS-v with adjuvant (Experimental): ISA-51-adjuvanted AGS-v emulsified in WFI (0.5mL)on Day 0 and on Day 21
  Interventions: Biological: AGS-v + adjuvant
- Placebo (Placebo Comparator): WFI (0.5mL) on Day 0 and Day 21
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AGS-v — AGS-v (unadjuvanted) as a suspension in WFI (0.5mL) on Day 0 and on Day 21
  Arms: AGS-v
Biological: AGS-v + adjuvant — ISA-51-adjuvanted AGS-v emulsified in WFI (0.5mL) on Day 0 and on Day 21
  Arms: AGS-v with adjuvant
Other: Placebo — WFI (0.5mL) on Day 0 and Day 21
  Arms: Placebo

SUMMARY:
Background:

Mosquitos carry diseases that cause major health problems and death worldwide. The AGS-v vaccine targets proteins in mosquito saliva. This may help prevent many mosquito-borne diseases. It might also reduce the lifespan of the mosquito that bites the vaccinated person.

Objective:

To see if the AGS-v vaccine is safe in humans and how it affects the immune system.

Eligibility:

Healthy adults ages 18-50

Design:

Participants will be screened another study.

Participants will be randomly assigned to get either the vaccine with a booster vaccine, the vaccine without the booster, or a placebo. These are given through a needle in the upper arm.

Participants will have visits that include medical history, physical exam, and blood and urine tests:

Baseline: They will get the vaccine and be monitored for 2 hours.

Follow-up visits 1 and 2 weeks after baseline.

Visit 3 weeks after baseline: They will get the booster and be monitored for 2 hours.

Follow-up visits 1 and 2 weeks after booster visit.

Visit 3-5 weeks after booster visit: This includes mosquito feeding. Mosquitos grown in the lab will be allowed to bite the arm. Blood will be drawn 4 times in the 3 hours after the feeding.

Phone follow-up a few days after the mosquito feeding.

After the feeding visit, 5 follow-up visits about every 2 months

Participants will keep a symptom diary for 7 days after each vaccine. They will record their temperature. They will measure any redness around the injection site. They will document and if possible photograph any mosquito bites they get.

DETAILED DESCRIPTION:
Mosquito-borne diseases continue to cause significant morbidity and mortality worldwide despite on-going control efforts. In 2015, there were >200 million cases of malaria worldwide, causing nearly half a million deaths, with most of the deaths occurring among children under the age of 5 years. Mosquitos also transmit arboviruses, including dengue, yellow fever, West Nile virus, chikungunya, Rift Valley fever, Japanese encephalitis, and Zika virus. The current new outbreak of Zika virus in Central and South America, as well as the Caribbean, serves as a reminder of how quickly these viruses can spread and how difficult they can be to control.

In this protocol we plan to perform a Phase I study of a novel universal mosquito-borne disease vaccine. Through modulation of the immune system after a mosquito feeding, this vaccine targets the vector saliva and may provide prophylaxis against multiple arboviral and protozoal diseases. In addition the vaccine potentially leads to a reduced mosquito lifespan after feeding therefore also reducing transmission of these diseases.

In this protocol we hope to demonstrate the safety of this vaccine similar to SEEK s other peptide based vaccines Flu-v and HIV-v that have been found to have very good safety profiles in previous Phase I trials. We also hope to demonstrate immunomodulation after a controlled clean Aedes aegypti mosquito feeding to demonstrate proof of concept efficacy of the vaccine. With the current rise of Zika in the Americas and the threat of local mosquito transmission in the U.S. and the rest of the world, a successful universal mosquito-borne disease vaccine offers the benefit of targeting this emerging disease as well as the many established infections such as dengue and malaria that make dealing with this newly emerging epidemic a challenge.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Healthy women and men who are greater than or equal to 18 and less than or equal to 50 years of age.
2. Willingness to complete all study visits and comply with all study requirements.
3. A male subject is eligible for the study if he agrees to practicing abstinence or using a condom with spermicide plus an acceptable form of contraception (see inclusion criteria 4) being used by any female partner from 4 weeks before study start to 12 weeks after the second vaccine administration.
4. A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

   * Of non-child bearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to study initiation through 12 weeks after the second vaccine administration. Acceptable methods of contraception include a male partner who is sterile and is the sole sexual partner of the female participant or a male partner who uses a condom with spermicide plus 1 or more of the following: 1) implants of levonorgestrel; 2) injectable progestogen; 3) an intrauterine device with a documented failure rate of <1%; 4) oral contraceptives; and 5) double barrier method including diaphragm.
5. Willing to have samples stored for future research (including genetic research).
6. Agrees to abstain from alcohol intake for 24 hours prior to each study visit.
7. Agrees to not donate blood or blood products throughout the study.

EXCLUSION CRITERIA:

1. Participant has any underlying or current medical condition, which, in the opinion of the Investigator, would interfere with the participation in the study.
2. Individual with body mass index (BMI) less than or equal to 18 and greater than or equal to 40.
3. Participants who have a clinically significant (as determined by the PI) baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table.
4. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
5. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
6. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
7. Self-reported or known history of alcoholism or drug abuse within 6 months prior to enrollment, or positive urine/serum test for drugs of abuse at screening
8. Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI to be a contraindication to protocol participation.
9. History of a previous severe allergic reaction with generalized urticaria, angioedema, anaphylaxis or anaphylactoid reaction.
10. Any condition or event that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent.
11. Has a known allergy to any of the components of the vaccine.
12. Has a history of severe immunization reaction.
13. Has a severe allergic reaction to mosquito bites

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Peng Z, Yang M, Simons FE. Immunologic mechanisms in mosquito allergy: correlation of skin reactions with specific IgE and IgG antibodies and lymphocyte proliferation response to mosquito antigens. Ann Allergy Asthma Immunol. 1996 Sep;77(3):238-44. doi: 10.1016/S1081-1206(10)63262-0. PMID 8814051
- [Background] Sidjanski S, Vanderberg JP. Delayed migration of Plasmodium sporozoites from the mosquito bite site to the blood. Am J Trop Med Hyg. 1997 Oct;57(4):426-9. doi: 10.4269/ajtmh.1997.57.426. PMID 9347958
- [Background] Ribeiro JM. Role of saliva in blood-feeding by arthropods. Annu Rev Entomol. 1987;32:463-78. doi: 10.1146/annurev.en.32.010187.002335. No abstract available. PMID 2880553
- [Derived] Manning JE, Oliveira F, Coutinho-Abreu IV, Herbert S, Meneses C, Kamhawi S, Baus HA, Han A, Czajkowski L, Rosas LA, Cervantes-Medina A, Athota R, Reed S, Mateja A, Hunsberger S, James E, Pleguezuelos O, Stoloff G, Valenzuela JG, Memoli MJ. Safety and immunogenicity of a mosquito saliva peptide-based vaccine: a randomised, placebo-controlled, double-blind, phase 1 trial. Lancet. 2020 Jun 27;395(10242):1998-2007. doi: 10.1016/S0140-6736(20)31048-5. Epub 2020 Jun 11. PMID 32534628

RESULTS

PARTICIPANT FLOW:
Groups:
- AGS-v: 825 µg (50 nmol each peptide) non-adjuvanted AGS-v vaccine 2 doses given 21 days apart
- AGS-v With Adjuvant: 825 µg (50 nmol each peptide) adjuvanted AGS-v vaccine 2 doses givemn 21 days apart
- Placebo: Placebo 2 doses given 21 days apart
Period: Overall Study
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Started | 16 | 17 | 16
Completed | 16 | 17 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AGS-v With Adjuvant: 825 µg (50 nmol each peptide) adjuvanted AGS-v vaccine 2 doses given 21 days apart
- Total: Total of all reporting groups
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 16 | 49
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 13 | 30
  Male | 7 | 9 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 2 | 10
  Not Hispanic or Latino | 13 | 12 | 14 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 8 | 18
  White | 9 | 8 | 6 | 23
  More than one race | 1 | 3 | 2 | 6
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: AEs Grade 3 or Higher
Description: Grade 3 or higher adverse events identified within 1 year after 2 vaccinations 21 days apart.
Time Frame: 1 year after vaccination (study duration)
Population: All subjects who received vaccination
Measure: Mean (95% Confidence Interval); unit: adverse events
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
adverse events | 0.44 [0.16 to 0.63] | 0.65 [0.23 to 0.93] | 0.63 [0.22 to 0.89]

2. Primary Outcome: GM-CSF Cytokine Level as Measured by Luminex
Description: Interferon-gamma and other cytokine markers of Th1 and Th2 response measured in vitro from PBMCs incubated with AGS-v antigens as indicators of Th1 vs. Th2 response
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1.106 (0.285) | 3.76 (6.05) | 1.101 (1.01)

3. Primary Outcome: IL-10 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 0.983 (0.048) | 1.088 (0.169) | 0.976 (0.055)

4. Primary Outcome: IL-1B Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1.009 (0.119) | 0.964 (0.105) | 0.946 (0.107)

5. Primary Outcome: IL-2 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1.173 (0.421) | 1.225 (0.372) | 1.115 (0.293)

6. Primary Outcome: IL-4 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1 (0.027) | 1.018 (0.047) | 0.991 (0.027)

7. Primary Outcome: IL-5 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1.267 (0.664) | 4.389 (13.32) | 1.022 (0.091)

8. Primary Outcome: Interferon-gamma Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 1.16 (0.568) | 1.613 (0.764) | 1.103 (0.307)

9. Primary Outcome: Number of Subjects With 1 or More Aes
Description: Percent of people with an AE
Time Frame: 1 year after vaccination (study duration)
Population: All subjects who received vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
Participants | 16 | 17 | 15

10. Primary Outcome: Number of Subjects With 1 or More Grade 3 or Higher AE
Description: Percent of people with a Grade 3 or higher AE
Time Frame: 1 year after vaccination (study duration)
Population: All subjects who received vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
Participants | 6 | 7 | 7

11. Primary Outcome: TNF-a Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
pg/mL | 0.995 (0.104) | 1.255 (0.573) | 0.993 (0.078)

12. Primary Outcome: Total AGS-v Specific Immunoglobulin
Description: Total AGS-v specific immunoglobulin measured in serum 14 days after the first and/or second vaccination.
Time Frame: 21 days after last vaccination
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 17 | 16
IU/mL | 0.9903 (0.373) | 4.3115 (5.08) | 1.0232 (1.42)

13. Secondary Outcome: GM-CSF Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 1.198 (1.289) | 1.8 (5.806) | 0.902 (0.296)

14. Secondary Outcome: IL-10 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 1.376 (2.029) | 1.749 (1.687) | 0.813 (0.206)

15. Secondary Outcome: IL-1B Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 0.905 (0.546) | 0.955 (0.281) | 0.758 (0.268)

16. Secondary Outcome: IL-2 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 1.027 (0.583) | 1.036 (0.138) | 0.98 (0.221)

17. Secondary Outcome: IL-4 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 1.034 (0.254) | 1.061 (0.157) | 0.915 (0.211)

18. Secondary Outcome: IL-5 Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 2.233 (4.085) | 3.113 (5.993) | 0.933 (0.119)

19. Secondary Outcome: Interferon-gamma Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 2.577 (3.954) | 2.004 (4.795) | 0.594 (0.792)

20. Secondary Outcome: Number of Adults Developed From 100 Eggs
Description: Measurement of changes to Aedes aegypti mosquito life cycle post feeding on blood from participants after vaccination
Time Frame: Day 42 Mosquito feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: Adult aedes aegypti mosquitoes
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Adult aedes aegypti mosquitoes | 69.13 (14.07) | 75.25 (13.55) | 78.53 (9.52)

21. Secondary Outcome: Number of Eggs Laid
Description: Measurement of changes to Aedes aegypti mosquito life cycle post feeding on blood from participants after vaccination
Time Frame: Day 42 Mosquito feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: Eggs
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Eggs | 706 (123.75) | 673.88 (221.29) | 663 (165.51)

22. Secondary Outcome: Number of Pupae Hatched of 100 Eggs
Description: Measurement of changes to Aedes aegypti mosquito life cycle post feeding on blood from participants after vaccination
Time Frame: Day 42 Mosquito feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: Number of hatched pupae
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Number of hatched pupae | 78.93 (13.08) | 79.62 (14.86) | 81.93 (9.08)

23. Secondary Outcome: Percent of Eggs That Developed Into Pupae
Description: Measurement of changes to Aedes aegypti mosquito life cycle post feeding on blood from participants after vaccination
Time Frame: Day 42 Mosquito feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: percentage of eggs
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
percentage of eggs | 11.59 (3.26) | 15.56 (13.58) | 13.76 (6.49)

24. Secondary Outcome: Percent of Pupae That Developed Into Adults
Description: Measurement of changes to Aedes aegypti mosquito life cycle post feeding on blood from participants after vaccination
Time Frame: Day 42 Mosquito feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: percentage of pupae
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
percentage of pupae | 88.12 (12.8) | 94.96 (6.86) | 95.77 (2.88)

25. Secondary Outcome: TNF-a Cytokine Level as Measured by Luminex
Description: as for outcome 2
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 15 | 12 | 12
pg/mL | 1.392 (3.464) | 1.382 (5.867) | 0.707 (0.554)

26. Secondary Outcome: Total AGS-v Specific Immunoglobulin
Description: Total AGS-v specific immunoglobulin measured in serum after the first and/or second vaccination.
Time Frame: 60 days after Day 42 Mosquito Feeding
Population: All subjects who received vaccination
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
Number analyzed (Participants) | 16 | 15 | 15
IU/mL | 1.0077 (0.29) | 3.6537 (4.45) | 1.2011 (1.27)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | AGS-v | AGS-v With Adjuvant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 16/16 | 17/17 | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGS-v (N=16) | AGS-v With Adjuvant (N=17) | Placebo (N=16)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Chills (General disorders) | 2 | 3 | 1
Fatigue (General disorders) | 5 | 8 | 4
Injection site erythema (General disorders) | 3 | 8 | 2
Injection site induration (General disorders) | 0 | 2 | 0
Injection site pain (General disorders) | 6 | 9 | 4
Injection site pruritus (General disorders) | 3 | 7 | 0
Injection site swelling (General disorders) | 2 | 9 | 1
Pyrexia (General disorders) | 1 | 7 | 4
Swelling (General disorders) | 15 | 16 | 15
Tenderness (General disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 5 | 7
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 2 | 1
Eosinophil count increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 8 | 6 | 5
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 3 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 2
White blood cell count increased (Investigations) | 2 | 1 | 1
White blood cells urine positive (Investigations) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 5
Headache (Nervous system disorders) | 7 | 8 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 15 | 15 | 15
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Systolic hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03055000/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT03055000/ICF_001.pdf